CLINICAL TRIAL: NCT06141148
Title: Clinical Presentaion, and Treatment Outcomes in Tuberculous Patients in Sohag Governorate
Brief Title: Clinical Presentation, and Treatment Outcomes in Tuberculous Patients in Sohag Governorate
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Mohamed Mohiedin Habeel, Resident-chest department-sohag hospital university, Sohag University
Other Study IDs: Soh-Med-23-10-012MS
Record Dates: First submitted 2023-11-15; First posted 2023-11-21 (Actual); Last update posted 2023-11-21 (Actual); Status verified 2023-11

CONDITIONS: Tuberculosis
MeSH Terms: conditions — Tuberculosis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- group A,: group A ( Pulmonary Tuberculosis).
  Interventions: Diagnostic Test: sputum analysis
- group B: group B ( Extra pulmnary Tuberculosis).
  Interventions: Diagnostic Test: lymph node biobsy

INTERVENTIONS:
Diagnostic Test: sputum analysis — sputum analysis to diagnose tuberculosis
  Groups: group A,
Diagnostic Test: lymph node biobsy — to diagnose tuberculous lymphadenitis
  Other Names: to diagnose tuberculous lymphadenitis
  Groups: group B

SUMMARY:
Tuberculosis (TB) is an infectious disease that commonly affects the lung and is caused by a bacterium called Mycobacterium Tuberculosis. The bacterium mostly affects people with impaired immunity TB becomes the second leading cause of morbidity and mortality among infectious diseases, following the emergence of the human immunodeficiency virus (HIV). HIV is the commonest risk factor for developing a life-threatening tuberculosis disease, on the other hand, HIV related immunodeficiency is worsened by TB infection.TB is among the top 10 causes of death worldwide. In2019, among 8.8 million adults who developed TB disease, 36% were women .TB has become the fifth leading cause of death among women.

ELIGIBILITY:
Inclusion Criteria:

* age above 18ys.
* confirmed diagnosis of tuberculosis.

Exclusion Criteria:

* childern.
* not confirmed diagnosis of tuberculosis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: * age above 18ys.
  * confirmed diagnosis of tuberculosis.
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2023-11-01 (Actual); Primary Completion 2024-12-30 (Estimated); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
percent of cured tuberculous patients | 1 year
  to detect percent of cured patients
percent of treatment failure | 1 year
  to detect percent of treatment failure in tuberculous patients

CONTACTS AND LOCATIONS:
Locations (1):
- Sohag university Hospital, Sohag, Egypt

REFERENCES:
- [Background] Ali MK, Karanja S, Karama M. Factors associated with tuberculosis treatment outcomes among tuberculosis patients attending tuberculosis treatment centres in 2016-2017 in Mogadishu, Somalia. Pan Afr Med J. 2017 Nov 2;28:197. doi: 10.11604/pamj.2017.28.197.13439. eCollection 2017. PMID 29610635
- [Background] Jalal TMT, Abdullah S, Wahab FA, Dir S, Naing NN. Prevalence and Factors Associated with Tuberculosis Treatment Success among TB/HIV Co-Infection in North-East Malaysia. Malays J Med Sci. 2017 Dec;24(6):75-82. doi: 10.21315/mjms2017.24.6.9. Epub 2017 Dec 29. PMID 29379389
- [Background] Mason PH, Snow K, Asugeni R, Massey PD, Viney K. Tuberculosis and gender in the Asia-Pacific region. Aust N Z J Public Health. 2017 Jun;41(3):227-229. doi: 10.1111/1753-6405.12619. Epub 2016 Dec 13. No abstract available. PMID 27960224
- [Background] Horton KC, MacPherson P, Houben RM, White RG, Corbett EL. Sex Differences in Tuberculosis Burden and Notifications in Low- and Middle-Income Countries: A Systematic Review and Meta-analysis. PLoS Med. 2016 Sep 6;13(9):e1002119. doi: 10.1371/journal.pmed.1002119. eCollection 2016 Sep. PMID 27598345